CLINICAL TRIAL: NCT03432559
Title: Local Side Effects of Transesophageal Echocardiography
Brief Title: Side Effects of Transesophageal Echocardiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ulrike Weber, Ass.Prof.Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 164/2009
Record Dates: First submitted 2018-02-01; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: endoscopy
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: endoscopy of pharynx, upper esophagus, mid esophagus, cardia, gastric fundus, and gastric body
Masking Description: the investigator doing the transesophageal examination will not be informed about the results of the endoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endoscopy (Other): endoscopy of the upper GI tract
  Interventions: Diagnostic Test: endoscopy

INTERVENTIONS:
Diagnostic Test: endoscopy — endoscopy of pharynx, upper esophagus, mid esophagus, cardia, gastric fundus, und gastric body

SUMMARY:
Transesophageal echocardiography is commonly used during cardiac surgery. Complications of transesophageal echocardiography are rare (1,2%), but are often underestimated and can lead to unrecognized blood loss and site of infection.

This study wants to assess the mucosa of pharynx, upper larynx, esophagus and stomach prior to and after echo probe insertion during cardiac surgery with endoscopy.

DETAILED DESCRIPTION:
Transesophageal echocardiography is commonly used during cardiac surgery. Main reasons for its use are the evaluation of cardiac function and valve morphology previous to and after cardiac surgery.

Complications of transesophageal echocardiography are rare (1,2%). Described complications may involve the gastrointestinal, cardiovascular or respiratory system.

The major complication of transesophageal echocardiography is local injury of the GI tract. Only massive bleeding and perforation were reported, minor injuries are not noticed in the early postoperative period but may play an important role, especially in patients discomfort, source of minor unrecognized blood loss and site of infection. As oropharyngeal bacteria are known to cause endocarditis and graft infection, this site of infection may be of special interest in cardiac surgery.

Study objectives:

To assess the mucosa of pharynx, upper larynx, esophagus and stomach prior to and after TEE probe insertion during cardiac surgery using flexible endoscopy.

Design:

Open, not randomized, observer blinded, pilot study. Inclusion criteria

* Planned cardiac surgery
* Age above 18 years
* Signed informed consent
* Clinical need for intraoperative use of transesophageal echocardiography Exclusion criteria
* Recent gastrointestinal pathologies (3-6 months)
* Recent operations of the upper gastrointestinal tract (3-6 months)
* Subjects not able to understand study procedures
* No signed informed consent
* Contraindications for transesophageal echocardiography

After induction of anesthesia and insertion of all needed catheters (arterial catheter, central venous catheter, bladder catheter, and pulmonary artery catheter, if indicated) an expert physician will perform the endoscopy (Olympus; Hamburg, Germany) of pharynx, esophagus, and stomach in order to exclude (respectively map) any alteration of the mucosa.

Immediately after endoscopy the transesophageal probe (6T, 6T-RS, 6Tc, 6Tc-RS Vivid GE; USA; X7-2T, S7-2omni, Philips), covered with a special condom, will be inserted. The TOE probe will remain 7-8 hours in the GI tract.

Two standard echocardiographic examinations are routinely performed during cardiac operation; the first (prior to skin incision) is assigned as baseline evaluation of cardiac morphology and function; the second (after weaning from cardiopulmonary bypass) is performed to check the result of the surgical procedure respectively to determine cardiac function for decision-making of medical treatment. A routine TEE - examination follows guidelines for standard TEE views and examination workflow and includes a minimum of 11 views up to a maximum of 28 views, depending on the type of pathology. Average time needed to perform a standard TEE examination varies from 5-15minutes.

For these reasons the number of TEE views per examination, the length of each examination, and the different probe positions (upper esophageal, mid esophageal, transgastric and deep transgastric) during examination and the length of stay of the probe in each position will be reported. As soon as the TEE probe has been removed the second endoscopy it will be performed in the same order as the baseline endoscopy.

Possible lesions of the mucosa will be classified as described by Geene et al. (Greene 1999, #9) as follows: erythema, edema, hematoma, mucosal erosion, petechiae, and perforation. In particular pharynx, upper esophagus, mid esophagus, cardia, gastric fundus, und gastric body will be examined.

The analysis of filmed examination will be performed by the endoscopist in a second time off-line, in a blind manner.

ELIGIBILITY:
Inclusion Criteria:

* Planned cardiac surgery
* Age above 18 years
* Signed informed consent
* Clinical need for intraoperative use of transesophageal echocardiography

Exclusion Criteria:

* Recent gastrointestinal pathologies (3-6 months)
* Recent operations of the upper gastrointestinal tract (3-6 months)
* Subjects not able to understand study procedures
* No signed informed consent
* Contraindications for transesophageal echocardiography
* Antibiotic treatment within three months prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2010-03-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
incidence of endoscopic mild mucosal injury | 7-8 hours
  erythema, edema, hematoma, mucosal erosion, petechiae, or perforation of the upper GI mucosa

SECONDARY OUTCOMES:
length of examination | 1 day
  Duration of the actual TEE examination
incidence of postoperative complications | up to 1 week
  GI bleeding, Perforation, swallowing difficulties

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Weber, M.D.Ph.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No